CLINICAL TRIAL: NCT00811668
Title: Crossover Comparison of Treatment With Continuous Positive Airway Pressure and Treatment With Adaptive Servo Ventilation (SOMNOventCR) in Patients With Underlying Heart Disease, Combined Obstructive Sleep Apnea and Cheyne-Stokes Respiration.
Brief Title: Comparison of CPAP With SOMNOventCR in Patients With Underlying Heart Disease, Combined OSA and CSR
Acronym: VCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: WI_VentCR_13/2008
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2011-08

CONDITIONS: Heart Diseases; Sleep Apnea, Central; Sleep Apnea, Obstructive
Keywords: Sleep Apnea Syndromes; heart diseases
MeSH Terms: conditions — Heart Diseases; Sleep Apnea, Central; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP before SOMNOVentCR (Experimental): started with CPAP and continued with SOMNOvent CR
  Interventions: Device: CPAP before SOMNOVentCR
- SOMNOVentCR before CPAP (Experimental): began with SOMNOvent CR and ended with CPAP
  Interventions: Device: SOMNOventCR before CPAP

INTERVENTIONS:
Device: CPAP before SOMNOVentCR — 4 weeks CPAP treatment, 1 week wash out period, 4 weeks SOMNOventCR treatment
  Arms: CPAP before SOMNOVentCR
Device: SOMNOventCR before CPAP — 4 weeks SOMNOventCR treatment, 1 week wash out period, 4 weeks CPAP treatment
  Arms: SOMNOVentCR before CPAP

SUMMARY:
In patients with underlying heart diseases like hypertensive heart disease, coronary heart disease or dilative cardiomyopathy obstructive sleep-apnea, central sleep-apnea and Cheyne-Stokes-respiration are common finding in polysomnography.

In a lot of these patients it is neither a purely obstructive sleep-apnea syndrome nor a complete Cheyne-Stokes-respiration but a combination of both sleep related respiratory disturbances.

Previous studies showed an improvement of the central respiratory disorder, for example Cheyne-Stokes-respiration, under continuous positive pressure breathing (CPAP) and an improvement of the left ventricular pump function. (Naughton 1995, Tkacova 1997).

However, the recently published CanPAP study could not prove any improvement in the mortality among CPAP therapy patients in comparison to the optimal medical treatment, although under this therapy, the number of breathing disturbances, the oxygen saturation at night and the ejection fraction of the left ventricle showed a significant improvement.(Bradley 2005)

Earlier studies proved the adaptive servo ventilation to be an effective therapy for patients with central sleep-apnea and Cheyne-Stokes-respiration respectively. (Teschler 2001) Teschler's study showed that the adaptive servo ventilation therapy with a reduction of central sleep apnea down to 10/hours succeeded. With the SOMNOvent CR a new therapy-algorithm has been developed for the adaptive servo ventilation in patients with obstructive sleep apnea and Cheyne-Stokes-respiration with underlying heart disease. In the first validation study this therapy was very effective and presented only few adverse effects in the patients. (Galetke 2007)

The goal of the study was to compare this new therapeutic option (SOMNOvent CR) with the established method of continuous positive airway pressure (CPAP) in patients with combination of obstructive sleep-apnea syndrome and Cheyne-Stokes-respiration with underlying heart disease.

DETAILED DESCRIPTION:
Patients who meet all the above mentioned criteria and who were diagnosed as sleep-apnoea syndrome patients in our hospital were asked to participate in the study.

We divided the patients in two groups:

Group 1: started with CPAP and continued with SOMNOvent CR Group 2: began with SOMNOvent CR and ended with CPAP

First of all a CPAP-titration was applied to both fixed groups during the second night. During the third night they received either the CPAP- pressure (first group) or the adaptive servo ventilation (second group. The patients were discharged from the hospital continuing with the procedure of the third night.

After four weeks a new admission for the sleep laboratory was necessary and, during the first night, a control investigation with the procedure of the last four weeks. The procedure changed during the next night, so that the patients of the first group now slept with the SOMNOventCR-device and the patients of the second group with the CPAP-device.

After a wash-out-period of a week and a four-week treatment with the last procedure a final in-hospital polysomnography was performed in which adaptive servo ventilation was applied to the first group and fixed CPAP to the second group.

After the study ended, the patients received the therapy procedure which was the most effective and which was better tolerated.

The following analyses were carried out in addition to the polysomnographic measurements:

Admission 1: Berlin questionnaire, European sleep questionnaire, echocardiography, 6 minute walking test, patients questionnaire.

Admission 2: ESS, Berlin questionnaire, echocardiography, 6 minute walking test, patients´ questionnaire.

After the wash-out-period: ESS, Berlin questionnaire, patients questionnaire.

Admission 4: ESS, Berlin questionnaire, echocardiography, 6 minute walking test, patients questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years.
* Diagnosis of arterial hypertension or a coronary heart disease or a dilative cardiomyopathy
* Combined sleep-apnea-syndrome with a total value of AHI>15 per hour and a rate up to 20% of central events or periodic breathing.

Exclusion Criteria:

* Heart failure NYHA-CLASS IV.
* Myocardial infarction or unstable angina pectoris or cardiac surgery within the last three months.
* Apnea-hypopnea-index < 15 per hour.
* Obstructive breathing disturbances up to 80%.
* Pregnancy.
* Absence of declaration of consent.
* Malign diseases.
* Serious (Severe) chronic oxygen-requiring pulmonary illness.
* Age under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
central apnea-hypopnea-index | February 2009

SECONDARY OUTCOMES:
Total apnea-hypopnea-index, minimum and mean oxygen saturation, compliance, subjective satisfaction with the therapy (questionnaire), left ventricular ejection fraction , six minutes walking distances. | February 2009

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Galetke, PD Dr., Study Chair; Winfried J. Randerath, Prof. Dr., Study Director

REFERENCES:
- [Background] Bradley TD, Logan AG, Kimoff RJ, Series F, Morrison D, Ferguson K, Belenkie I, Pfeifer M, Fleetham J, Hanly P, Smilovitch M, Tomlinson G, Floras JS; CANPAP Investigators. Continuous positive airway pressure for central sleep apnea and heart failure. N Engl J Med. 2005 Nov 10;353(19):2025-33. doi: 10.1056/NEJMoa051001. PMID 16282177
- [Background] Naughton MT, Liu PP, Bernard DC, Goldstein RS, Bradley TD. Treatment of congestive heart failure and Cheyne-Stokes respiration during sleep by continuous positive airway pressure. Am J Respir Crit Care Med. 1995 Jan;151(1):92-7. doi: 10.1164/ajrccm.151.1.7812579.
- [Background] Teschler H, Dohring J, Wang YM, Berthon-Jones M. Adaptive pressure support servo-ventilation: a novel treatment for Cheyne-Stokes respiration in heart failure. Am J Respir Crit Care Med. 2001 Aug 15;164(4):614-9. doi: 10.1164/ajrccm.164.4.9908114. PMID 11520725
- [Background] Tkacova R, Hall MJ, Liu PP, Fitzgerald FS, Bradley TD. Left ventricular volume in patients with heart failure and Cheyne-Stokes respiration during sleep. Am J Respir Crit Care Med. 1997 Nov;156(5):1549-55. doi: 10.1164/ajrccm.156.5.9612101. PMID 9372674
- [Background] Javaheri S, Parker TJ, Liming JD, Corbett WS, Nishiyama H, Wexler L, Roselle GA. Sleep apnea in 81 ambulatory male patients with stable heart failure. Types and their prevalences, consequences, and presentations. Circulation. 1998 Jun 2;97(21):2154-9. doi: 10.1161/01.cir.97.21.2154. PMID 9626176